CLINICAL TRIAL: NCT01855464
Title: Pulmonary Wedge Resection Plus Parietal Pleurectomy (WRPP) Versus Parietal Pleurectomy (PP) for the Treatment of Recurrent Primary Pneumothorax
Brief Title: Wedge Resection or Parietal Pleurectomy for the Treatment of Recurrent Pneumothorax (WOPP)
Acronym: WOPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Otto-von-Guericke University Magdeburg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Torsten Walles, Univ. Prof. Dr. med. Thorsten Walles, Director, thoracic surgery, Otto-von-Guericke University Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKW-TCH-2013-001; German Research Foundation (Other Grant/Funding Number: DFG WA 1649/5-1)
Record Dates: First submitted 2013-05-06; First posted 2013-05-16 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Pneumothorax; Recurrent Pneumothorax
Keywords: pneumothorax; primary pneumothorax; lung collapse
MeSH Terms: conditions — Pneumothorax; Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wedge resection+parietal pleurectomy (Experimental): Surgical treatment includes parietal pleurectomy and wedge resection of the tip of the lung.
  Interventions: Procedure: wedge resection; Procedure: parietal pleurectomy
- parietal pleurectomy (Active Comparator): Surgical therapy is limited to parietal pleurectomy.
  Interventions: Procedure: parietal pleurectomy

INTERVENTIONS:
Procedure: wedge resection — Complementary to parietal pleurectomy lung tissue is resected.
  Arms: wedge resection+parietal pleurectomy
Procedure: parietal pleurectomy — The parietal pleura is resected for treating primary pneumothorax.

SUMMARY:
Primary spontaneous pneumothoraces (PSP) represent a significant public health problem, occurring in young healthy subjects without pre-existing lung disease or precedent medical intervention or trauma with a reported incidence of up to 18-28/100 000 per year. PSP treatment often requires thoracic surgery to restore lung expansion and to prevent de novo lung collapse. Despite the presence of elaborated guidelines by the British Thoracic Society (BTS) postulating apical wedge resection of the lung and total parietal pleurectomy (WRPP), the majority of German hospitals gathered experience especially in limiting surgery to cost-saving partial apical parietal pleurectomy or yet apical pleural abrasion (PP). Until today, hardly any reliable data exist to analyze and compare the varying treatment approaches regarding efficacy and efficiency. In this randomized, multi-centric clinical trial, both treatment approaches will be compared. For this purpose, candidates for surgery will be randomized into one of the two treatment groups after informed consent has been obtained. Patients will be followed for 2 years by the participating centres to be able to evaluate the long-term effect of the surgical interventions.

DETAILED DESCRIPTION:
The trial will be conducted at the major thoracic surgery units in Germany. Each centre can include patients on the basis of the presence of a PSP and the inclusion and exclusion criteria.

After informed consent has been obtained from the study participants, each has to fill out the standardized short-form health survey (SF-36) questionnaire and the visual analogue scale (VAS) to determine baseline parameters for the (current) state of health and pain level.Randomization into the two interventional groups is carried out before surgery.

Patients are operated according to good clinical practice either by pleurectomy alone (PP) or total parietal pleurectomy with apical wedge resection of the pulmonary apex (WRPP). Procedure related parameters (like operation time, applied suture materials including staplers) are documented.

The postoperative care is subject to each participating centre's standards. The postoperative course is evaluated (mortality, morbidity, duration of tube drainage, re-interventions or operations, length of stay, need for blood substitutions).

To evaluate the long term effect of the surgical intervention, all study participants are followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* recurrence of a primary pneumothorax
* persistent primary pneumothorax
* patient preference (in primary events)

Exclusion Criteria:

* presence of a pulmonal fistula
* underlying lung disease
* previous thoracic surgery (except tube thoracostomy)
* previous pleurodesis
* conversion thoracotomy

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-11; Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of primary pneumothorax following VAT surgery | 2 years
  Patients are followed to identify all incidents of recurrent lung collapse following VAT surgery. Suspected recurrences will be confirmed by chest X-ray.

SECONDARY OUTCOMES:
postoperative morbidity | 30 days
  postoperative complications
postoperative pain | 7 days
  rest and stress with a pain scale ranging from 1 to 10 (measured with the Visual Analogue Scale - VAS)
function quality of life | 2 years
  measured with SF-36 Health Survey (The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability Sections:Vitality;Physical functioning;Bodily pain;General health perceptions;Physical role functioning;Emotional role functioning;Social role functioning;Mental Health)
costs of treatment | up to 30 days
  documentation of postoperative Hospitalization, the number of trocars

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Walles, MD, Study Chair — Magdeburg University Hospital
Locations (23):
- Germany (23):
  - Klinikum rechts der Isar München, München, Bavaria
  - Universitätsklinikum Magdeburg A. ö. R., Magdeburg, Saxony-Anhalt
  - Charité, Berlin
  - Vivantes Thoraxzentrum, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - DRK Kliniken Berlin, Berlin
  - Lungenklinik Köln Merheim, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - LungenClinic Grosshansdorf, Großhansdorf
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg-Eppendorf
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Asklepios Klinik Langen, Langen
  - LMU München, München
  - Asklepios Fachklinik, München-Gauting
  - Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - Robert Bosch Krankenhaus, Stuttgart
  - Johanniter-Krankenhaus im Fläming Treuenbrietzen GmbH, Treuenbrietzen
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry M, Arnold T, Harvey J; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of spontaneous pneumothorax. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii39-52. doi: 10.1136/thorax.58.suppl_2.ii39. No abstract available. PMID 12728149
- [Background] Chan JW, Ko FW, Ng CK, Yeung AW, Yee WK, So LK, Lam B, Wong MM, Choo KL, Ho AS, Tse PY, Fung SL, Lo CK, Yu WC. Management of patients admitted with pneumothorax: a multi-centre study of the practice and outcomes in Hong Kong. Hong Kong Med J. 2009 Dec;15(6):427-33. PMID 19966346
- [Background] Gossot D, Galetta D, Stern JB, Debrosse D, Caliandro R, Girard P, Grunenwald D. Results of thoracoscopic pleural abrasion for primary spontaneous pneumothorax. Surg Endosc. 2004 Mar;18(3):466-71. doi: 10.1007/s00464-003-9067-z. Epub 2004 Feb 2. PMID 14752638
- [Derived] Neudecker J, Malzahn U, Heuschmann P, Behrens U, Walles T. Pulmonary wedge resection plus parietal pleurectomy (WRPP) versus parietal pleurectomy (PP) for the treatment of recurrent primary pneumothorax (WOPP trial): study protocol for a randomized controlled trial. Trials. 2015 Nov 30;16:540. doi: 10.1186/s13063-015-1060-z. PMID 26620271
- See also: Click here for information on German Research Foundation Grant — http://gepris.dfg.de/gepris/OCTOPUS/;jsessionid=E6A2D8650C043C03A91FE2EC2CE5C091?context=projekt&id=209750507&module=gepris&task=showDetail
- See also: Official Trial Website — http://www.wopp-studie.de